CLINICAL TRIAL: NCT02331927
Title: Personalized Marker-driven Early Switch to Aflibercept in Patients With Metastatic Colorectal Cancer (PERMAD-Trial) - a Multicenter, Multinational, Two Part, Phase II Trial
Brief Title: PERMAD: Personalized Marker-driven Early Switch to Aflibercept in Patients With Metastatic Colorectal Cancer
Acronym: PERMAD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Ulm (Other)
Collaborators: Hubertus-Wald-Cancer Center Hamburg, Germany (Unknown); Sanofi (Industry); Assign Data Management and Biostatistics GmbH (Other)
Responsible Party: Principal Investigator, Thomas Seufferlein, Prof. Dr. Thomas Seufferlein, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PERMAD; 2012-005657-24 (EudraCT Number)
Record Dates: First submitted 2014-09-10; First posted 2015-01-06 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer; marker-driven; bevacizumab; aflibercept; cytokines; angiogenic factors; CAF
MeSH Terms: conditions — Colorectal Neoplasms | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Randomized Part: Arm A (No Intervention): Conventional switch of chemotherapy together with the antiangiogenic treatment: Bevacizumab and mFOLFOX6 (continuation of same regimen until progressive disease (PD) according to RECIST v1.1, followed by switch to aflibercept and FOLFIRI after PD).
- Ramdomized Part: Arm B (Experimental): Early marker-driven switch of anti-angiogenic agent and maintenance of chemotherapy: Bevacizumab and mFOLFOX6 will be administered until change of the CAF-profile and at least stable disease according to RECIST v1.1. Change to Aflibercept and mFOLFOX6 (change of bevacizumab to aflibercept and continuation of mFOLFOX6) until PD according to RECIST v1.1, followed by change to FOLFIRI after PD).
  Interventions: Biological: Aflibercept

INTERVENTIONS:
Biological: Aflibercept — Early marker-driven switch of antiangiogenic treatment (bevacizumab to aflibercept) maintaining the chemotherapy backbone until definite radiological progression.
  compared to a conventional treatment approach of changing chemotherapy and antiangiogenic agent at time of radiologic progression.
  Arms: Ramdomized Part: Arm B

SUMMARY:
The primary objective of the two phase PERMAD trial is the evaluation of the impact of a personalized marker-driven treatment approach with early detection of progression and modification of treatment on cytokines and angiogenic factors (CAF) and efficacy.

In regard of the two parts, the primary objective of the run-in phase (n=50 patients) with conventional switch of chemotherapy together with the anti-angiogenic agent is the determination of a distinct cytokines and angiogenic factor (CAF) profile during treatment with FOLFOX and bevacizumab, which allows early detection/prediction of progressive disease. The primary objective of the marker-driven randomized part (n=150 patients) with marker-driven switch of antiangiogenic agent and maintenance of chemotherapy is the evaluation of the efficacy of an early marker-driven switch of anti-angiogenic treatment (bevacizumab to aflibercept)

This is a multicentre, multinational, open labeled, prospective, randomized, controlled phase II study designed to assess the clinical utility of an early marker driven change of anti-angiogenic treatment (bevacizumab to aflibercept) maintaining the chemotherapy backbone until definite radiological progression in first line treatment of patients with metastatic colorectal cancer. After completing the run in phase of the study, with at least 30 patients completing their first line treatment (due to progression, secondary resection or toxicity) and being evaluable for CAF analyses, the results will be reviewed by an Independent Data Monitoring Committee (IDMC). Based on that review the decision to continue with, modify or cancel the randomized part will be made.

The primary endpoint of the run-in phase with conventional switch of chemotherapy together with the anti-angiogenic agent is:

• Progression free survival (PFS1) of first line treatment

The primary endpoint of the randomized part with marker-driven switch of antiangiogenic agent and maintenance of chemotherapy is:

• Progression free survival rate at 6 months (PFSR@6) after first cycle after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of colorectal cancer presenting with unresectable stage IV (UICC) disease (primary tumor may be present)
* Patients with at least one measurable lesion, with size > 1 cm (RECIST v1.1)
* ECOG Performance status ≤ 2
* Life expectancy > 3 months
* Age ≥18 years.
* Haematologic function: ANC ≥ 1.5 x 109/L, platelets ≥ 100 x109/L, hemoglobin ≥ 9 g/dl or 5.59 mmol/l
* Patients not receiving therapeutic anticoagulation must have an INR < 1.5 and aPTT < 1.5 x ULN within 7 days prior to enrollment. The use of full dose anticoagulants is allowed as long as the INR or aPTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose for anticoagulants for at least two weeks at the time of enrollment.
* Adequate liver function as measured by serum transaminases (AST & ALT) ≤ 2.5 x ULN (in case of liver metastases < 5 x ULN) and total bilirubin ≤ 1.5 x ULN
* Adequate renal function: Serum creatinine ≤ 1.5 x ULN
* Signed, written informed consent
* At least 6 months after completion of adjuvant chemotherapy.

Exclusion Criteria:

* Treatment with any other investigational agent within 30 days prior to entering this study.
* Prior systemic or local treatment of metastatic disease.
* Prior adjuvant or neo-adjuvant chemotherapy/radiotherapy completed less than 6 months prior to study entry.
* Pre History or evidence upon physical/neurological examination of CNS disease (unrelated to cancer) (unless adequately treated with standard medical therapy) e.g. uncontrolled seizures.
* Fertile women (< 1 year after last menstruation) and men of childbearing potential unwilling or unable to use effective means of contraception (adequate: intrauterine device, long-acting injection, hormon implant, vasectomy) during treatment and for 6 months after the end of treatment.
* Pregnancy or lactation
* Positive serum pregnancy test within 7 days of starting study treatment in premenopausal women and women < 1 year after the onset of menopause.
* Past or current history (within the last 2 years prior to treatment start) of other malignancies except metastatic colorectal cancer (patients with curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible).
* Peripheral neuropathy NCI CTCAE-grade ≥ 1
* Known DPD-insufficiency.
* Active inflammatory bowel disease or other bowel disease causing chronic diarrhea (defined as > 4 loose stools per day)
* History of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis) haemoptoe or evidence of interstitial lung disease on baseline CT scan.
* Serious, non-healing wound, ulcer or bone fracture.
* Thrombosis or severe bleeding within 6 months prior to entry into the study (except for bleeding of the tumor before its surgical resection) and no evidence of bleeding diathesis or coagulopathy.
* Urine dipstick for proteinuria ≥ 2+. If urine dipstick is ≥ 2+, 24-hour urine must demonstrate ≤ 1 g of protein in 24 hours for patient to be eligible.
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to treatment.
* Clinically significant cardiovascular disease, for example CVA, myocardial infarction (≤ 12 months before treatment start), unstable angina, NYHA Class II CHF, arrhythmia requiring medication, or uncontrolled hypertension.
* Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.
* Known hypersensitivity or contraindication to the drugs used in the trial (eg: aflibercept, 5-FU, folinic acid/ leucovorin, oxaliplatin, bevacizumab, irinotecan).
* Concomitant treatment with ASS > 325 mg/d or NSAIDs, known to inhibit platelet function, sorivudin or analog compounds or preparations of St. John's wort.
* Inability or unwillingness to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-03; Primary Completion 2020-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Run-in phase: Progression free survival (PFS1) of first line treatment | approx. 10-12 months
  Run-in phase with conventional switch of chemotherapy together with the anti-angiogenic agent.
  Primary endpoint:
  • Progression free survival (PFS1) of first line treatment Randomized part with marker-driven switch of antiangiogenic agent and maintenance of chemotherapy.
  Primary endpoint:
  • PFS rate at 6 months (PFSR@6) after first cycle after randomization
Randomized part: PFS rate at 6 months after first cycle after randomization | 6 months
  Randomized part with marker-driven switch of anti-angiogenic treatment

SECONDARY OUTCOMES:
Predictive value of CAF particularly PlGF and VEGF-B for early detection of progression during treatment with chemotherapy and bevacizumab | approx. 10-12 months
Determination and validation of a CAF profile based on PlGF and VEGF-B predicting tumor progression before radiologic progression | approx. 10-12 months
PFS1, after first cycle after randomization (PFSr) and of second line treatment (PFS2) | approx. 20 months
Time to randomization (TTR) | approx. 10-12 months
Overall survival (OS) | 5 years
Overall response rate (RR) and Secondary resection rate (sRR) | approx. 20 months
Toxicity, Quality of life (QoL) | approx. 20 months
Changes in CAF during early marker-driven switch and conventional treatment approach | approx. 20 months
Prognostic value of CAF at baseline and/or during treatment | approx. 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Seufferlein, Prof. Dr., Principal Investigator — University of Ulm
Locations (3):
- Germany (3):
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Klinikum am Steinenberg Reutlingen, Reutlingen
  - University of Ulm, Ulm